CLINICAL TRIAL: NCT01988831
Title: Phase 2 Prospective Study of the Efficacy of Propranolol on Malignant Melanoma Progression. A Randomized Placebo-controlled,Single Blind Trial
Brief Title: Efficacy of Propranolol Treatment to Prevent Melanoma Progression
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: We must delay the study for some financial reasons
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Le Gal, Associate Physician, PD, MD/PhD, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUG-MEL-BB
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Stages III Skin Melanoma; Stages II Skin Melanoma; Stage IB Skin Melanoma
Keywords: Malignant melanoma; betablocker; propranolol; interventional; prospective; adjuvant; recurrence
MeSH Terms: conditions — Melanoma; Recurrence | interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 113 patients will be enrolled in the placebo group with respect to randomization.
  Placebo group will be prescribed placebo pills in the same packaging as propranolol treated group.
  The frequency and duration of the treatment is the same as propranolol arm. The placebo group will have the same cardiology consultation as propranolol treated group to ensure the respect of blindness.
  Interventions: Drug: Placebo pill
- Betablocker (Experimental): drug: 'Propranolol hydrochloride' 338 patients will be enrolled in the "Propranolol" Group and treated with propranolol.
  The dosage will be determined by the cardiologist as the maximum tolerated dose to a maximum of 160mg/day.
  One long acting pill a day until an evidence of disease progression or the end of the study.
  Interventions: Drug: Propranolol hydrochloride

INTERVENTIONS:
Drug: Propranolol hydrochloride — This intervention apply to Propranolol group
  Other Names: Inderal; Avlocardyl; Hemipralon LP; Propranolol EG; PROPRANOLOL Ratiopharm; Propranolol Teva
  Arms: Betablocker
Drug: Placebo pill — We use placebo pills alike propranolol commercial pills to ensure blindness of the subjects during the study.
  Arms: Placebo

SUMMARY:
Melanoma's incidence is increasing worldwide. The efforts made in melanoma screening led to an earlier detection of the primary tumour and a better prognosis, but melanoma remains an aggressive cancer when it comes to its metastatic stage. Three recent retrospective studies compared groups of patients diagnosed with primary melanoma and treated with betablockers for another indication to patients who never received betablockers. In these three studies, the outcome of the disease is significantly better for people under betablocker treatment with a decreased rate of recurrence and a better 5 years survival rate. Here we want to investigate the efficacy and the tolerability of an adjuvant treatment with propranolol for patients suffering from a primary melanoma with a high risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 y.o
* Breslow index > 1mm or any Breslow index with ulcerated primary lesion
* Melanoma stage AJCC Ib, IIa, IIb, IIc, IIIa, IIIb or IIIc
* Able to undergo outpatient treatment

Exclusion Criteria:

* No contra indication for betablockers as defined by the compendium
* No clinical evidence of coagulopathy
* No unstable angina pectoris
* No AV-block II or III without pacemaker
* No severe congestive heart failure
* No untreated phaeochromocytoma
* No severe bradycardia
* No severe hypotension
* No severe impairment of peripheral arterial circulation
* No uncontrolled cardiac arrhythmia
* No severe asthma or COPD
* No uncontrolled diabetes mellitus
* No Angioneurotic edema
* No severe Aortic valve stenosis
* No severe hypertrophic cardiomyopathy
* No severe renal dysfunction
* No patients on beta blockers by inclusion
* No known adverse reaction to betablockers
* No pregnant or lactating patients can be included
* No melanoma stage AJCC IV by inclusion
* No patients requiring a specific oncological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2016-06; Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of propranolol on progression free survival for patients suffering from a primary melanoma with a high risk of recurrence | five years
  The efficacy of propranolol treatment will be tested in one interim analysis when the last patient enrolled have reached one year of follow up and one final analysis when the last patient enrolled have reached three years of follow up. The primary endpoint of the study will be the progression of the disease.
  We will measure the efficacy of a propranolol treatment on the risk of progression of the disease.

SECONDARY OUTCOMES:
Use of serum microRNA profile as a predictor for recurrence | 5 years
  We will investigate the microRNA profile in the serum of patients of both groups during the whole study to identify biomarkers specific for recurrence.
Overall survival | 5 years
  We investigate the impact of propranolol treatment on the 5 years survival.

CONTACTS AND LOCATIONS:
Overall Officials: Frédérique-Anne Le Gal, MD/PhD, Principal Investigator — Hôpital cantonal universitaire de Genève
Locations (1):
- Hôpital universitaire de Genève, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Background] De Giorgi V, Grazzini M, Gandini S, Benemei S, Lotti T, Marchionni N, Geppetti P. Treatment with beta-blockers and reduced disease progression in patients with thick melanoma. Arch Intern Med. 2011 Apr 25;171(8):779-81. doi: 10.1001/archinternmed.2011.131. PMID 21518948
- [Background] Lemeshow S, Sorensen HT, Phillips G, Yang EV, Antonsen S, Riis AH, Lesinski GB, Jackson R, Glaser R. beta-Blockers and survival among Danish patients with malignant melanoma: a population-based cohort study. Cancer Epidemiol Biomarkers Prev. 2011 Oct;20(10):2273-9. doi: 10.1158/1055-9965.EPI-11-0249. Epub 2011 Sep 20. PMID 21933972
- [Background] De Giorgi V, Gandini S, Grazzini M, Benemei S, Marchionni N, Geppetti P. Effect of beta-blockers and other antihypertensive drugs on the risk of melanoma recurrence and death. Mayo Clin Proc. 2013 Nov;88(11):1196-203. doi: 10.1016/j.mayocp.2013.09.001. PMID 24182700